CLINICAL TRIAL: NCT03479372
Title: A Randomized, Double Masked, Uncontrolled , Multicenter Phase I/II Study to Evaluate Safety and Tolerability of PAN-90806 Eye Drops, Suspension in Treatment-Naïve Participants With Neovascular Age-Related Macular Degeneration (AMD)
Brief Title: Study of PAN-90806 Eye Drops, Suspension for Neovascular AMD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PanOptica, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PAN-01-102
Record Dates: First submitted 2018-03-14; First posted 2018-03-27 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: AMD; wet AMD; exudative AMD; macular degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking will be maintained by using a coded drug supply.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- PAN-90806 Eye Drops, dose 1 (Experimental): PAN-90806 Ophthalmic Suspension taken once daily for 12 weeks
  Interventions: Drug: PAN-90806 Ophthalmic Suspension
- PAN-90806 Eye Drops, dose 2 (Experimental): PAN-90806 Ophthalmic Suspension taken once daily for 12 weeks
  Interventions: Drug: PAN-90806 Ophthalmic Suspension
- PAN-90806 Eye Drops, dose 3 (Experimental): PAN-90806 Ophthalmic Suspension taken once daily for 12 weeks
  Interventions: Drug: PAN-90806 Ophthalmic Suspension

INTERVENTIONS:
Drug: PAN-90806 Ophthalmic Suspension — PAN-90806 provided in single-use dropper bottles for topical ocular administration
  Other Names: PAN-90806 Eye Drops

SUMMARY:
Double-masked, uncontrolled, multi-center, study in which participants will be randomized to one of 3 doses of topical ocular PAN 90806 administered once daily for 12 weeks.

DETAILED DESCRIPTION:
Patients with newly diagnosed, active, pathologic CNV associated with neovascular AMD will be screened for inclusion into the study after providing written informed consent. Participants who are eligible for the study will be centrally randomized at Day 1 to one of three doses of PAN-90806 Eye Drops. Participants will be instructed to apply one drop of PAN-90806 to the ocular surface of the identified study eye once daily for twelve (12) weeks.

Participants will return for follow-up visits at Week 2, Week 4, Week 8, Week 12, 1 week after stopping PAN-90806 treatment and 1 month after stopping PAN-90806 treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis in the study eye of active, pathologic, newly diagnosed and previously untreated, subfoveal choroidal neovascular (CNV) lesions secondary to neovascular AMD
* Aged 50 years or older
* Demonstrate the ability, or have a family member who is willing and able, to instill topical ocular drops in the study eye

Exclusion Criteria:

* Prior ocular or systemic treatment or surgery for neovascular AMD in the study eye
* Prior use within the last 3 months or a high possibility of requiring treatment with anti-VEGF therapy in the fellow eye during the study
* Significant retinal serous pigment epithelial detachment (PED), atrophy, or fibrosis/scar involving the fovea
* History of or current clinical evidence in the study eye of aphakia, diabetic macular edema, any ocular inflammation or infections, pathological myopia, retinal detachment, advanced glaucoma, and/or significant media opacity, including cataract
* History or evidence of the following surgeries in the study eye: penetrating keratoplasty or vitrectomy; corneal transplant; corneal or intraocular surgery within 3 months of Screening
* Uncontrolled hypertension despite use of antihypertensive medications
* Participation in any investigational drug or device study, systemic or ocular, within past 3 months
* Women who are pregnant or nursing
* Women of child-bearing potential who are not using a highly effective form of birth control
* Known serious allergies or hypersensitivity to the fluorescein dye used in angiography or to the components of the PAN-90806 formulation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2019-05-27 (Actual); Study Completion 2019-06-27 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events | up to 12 weeks

SECONDARY OUTCOMES:
Mean change from baseline in study eye ETDRS Visual Acuity | through Week 12
Mean change from baseline in study eye retinal thickness | through Week 12
Number of patients needing additional treatment with ranibizumab | through Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Martin Wax, MD, Study Director — PanOptica, Inc.
Locations (18):
- United States (8):
  - Colorado Retina Associates, Golden, Colorado
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Retinal Consultants of Nevada, Henderson, Nevada
  - Retinal Consultants of Nevada, Las Vegas, Nevada
  - Retina Center of New Jersey, Bloomfield, New Jersey
  - Retina Center of New Jersey, Teaneck, New Jersey
  - Vision Research Center, Albuquerque, New Mexico
  - Duke University, Durham, North Carolina
- Czechia (2):
  - Fakultní nemocnice Královské Vinohrady, Prague
  - Axon Clinical, Prague
- Hungary (2):
  - Semmelweis University, Budapest
  - University of Debrecen, Debrecen
- P. Stradina Clinical University hospital, Riga, Latvia
- United Kingdom (5):
  - Barnet Hospital, Barnet, Hertfordshire
  - New Cross Hospital, Wolverhampton, West Midlands
  - Bradford Royal Infirmary, Bradford
  - Moorefields Eye Hospital, London
  - Manchester Royal Eye Hospital, Manchester